CLINICAL TRIAL: NCT03510416
Title: Efficacy and Safety of Apatinib Combined With TACE in Patients With Hepatocellular Carcinoma Refractory to Transcatheter Arterial Chemoembolization
Brief Title: Efficacy and Safety of Apatinib Combined With TACE in Patients With Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-IR-2018
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma Refractory to Transcatheter Arterial Chemoembolization
Keywords: apatinib，TACE， hepatocellular carcinoma
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib combined with TACE (Experimental): Apatinib is administered after TACE 4-7 days, and TACE treatment is performed after discontinuation of apatinib for 4 days.Every 28 days is a cycle.
  Interventions: Drug: Apatinib; Radiation: TACE

INTERVENTIONS:
Drug: Apatinib — apatinib is a kind of Inhibitor of VEGFR-2
Radiation: TACE — Epirubicin,ultra-fluid lipiodol and gelatin sponge articles are used in TACE.

SUMMARY:
Efficacy and Safety of Apatinib Combined With TACE in Patients With Hepatocellular Carcinoma Refractory to Transcatheter Arterial Chemoembolization .

DETAILED DESCRIPTION:
Aptinib combined with TACE can be generated through embolization and angiogenesis by the dual target of vascular suppression.Efficacy and safety of apatinib combined with TACE in patients with hepatocellular carcinoma refractory to transcatheter arterial chemoembolization.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old;Estimated survival time≥12 weeks
* Histologicaly and cytologicaly diagnosed as Hepatocellular carcinoma of the liver ( HCC ) and with At least one imaging examination of measurable lesions (RECIST), CT or MR scan Long diameter of tumor ≥ 10 mm.Target lesion without Local treatment
* Child-pugh liver function Rating: A level, B level
* BCLC Staging as B / C period
* ECOG 0-1
* Have progressed after at least twice TACE
* The main organ function is normal, and meet the following standards:(1)The standard of blood routine examination should be consistent: HB≥90 g/L, ANC≥1.5×10^9/L, PLT≥60×10^9/L; (2)Biochemical tests should meet the following criteria: ALB ≥29 g/L；TBIL<2'ULN, ALT and AST<5'ULN,Cr ≤ 1.5*ULN
* Fertile woman must perform a pregnancy test (serum or urine) 7 days before screened, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib. For man, surgical sterilization should be performed, or voluntarily adopt proper methods of contraception during the observation period and 8 week after the last given apatinib
* Patients voluntarily entered the study and signed informed consent form (ICF).

Exclusion Criteria:

* Received Any local treatment other than TACE (including but not limited to surgery, radiotherapy, hepatic arterial embolization, hepatic arterial infusion, radiofrequency ablation, cryoablation, or percutaneous ethanol injection) within four weeks before randomization
* Participated in other cancer drug clinical trials within four weeks before randomization
* hepatobiliary cell carcinoma and mixed cell carcinoma are known; previous ( 5 year) or at the same time suffering from other incurable malignancies, except for the cured basal cell carcinoma of the skin and cervical carcinoma in situ
* have received or Prepared for liver transplantation
* A serous cavity effusion (including hydrothorax, ascites, pericardial effusion) with local symptoms requiring local treatment; or Child-Pugh>2；
* Patients with uncontrol hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg, despite optimal drug therapy)
* Suffering from coronary heart disease, arrhythmia or grade II (including QTc prolongation > 450 ms male, female, 470 MS) and Cardiac insufficiency
* According to NYHA standard, III ~ IV cardiac insufficiency, or heart colour to exceed revealed left ventricular ejection fraction (LVEF) < 50%
* There are several factors that affect oral medicine,such as unable to swallow, chronic diarrhea and intestinal obstruction
* Before randomization within 6 months had significant bleeding clinical significance or definite bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, baseline fecal occult blood and above, or suffering from vasculitis
* History of abdominal fistula, gastrointestinal perforation or abdominal abscess within 28 days before randomization
* Abnormal coagulation (INR>1.5 or PT>ULN+4, or APTT>1.5 ULN), bleeding tendency or receiving coagulation therapy
* Central nervous system with symptoms of metastasis
* there is typical interstitial pneumonia or pulmonary fibrosis
* Patients with a history of psychiatric drug abuse and can not be prevented or have mental disorders
* before participating in the study 7 days use strong-effect in CYP3A4 inhibitor therapy, or prior to participating in the study 12 days use the strong-effect in CYP3A4 inducer Therapy
* pregnant or lactating women who are not willing or unable to take effective contraceptive measures
* A history of mental illness, or psychotropic substance abuse
* Patients with allergies to research drugs
* Other patients who were considered unsuitable for inclusion by physicians.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time To Progression | From the date of first procedure of apatinib combined with TACE until the time when the disease progresses, assessed up to 14 months
  Time to progression is defined as stable with treatment of apatinib combined with TACE after enrollment until lesions are defined as disease progression.

SECONDARY OUTCOMES:
Overall Survival | From the date of randomization until the date of death from any cause, assessed up to 14 months
  From the date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: zhiping Yan, MD, Study Director — Department of Interventional Radiology, Zhongshan Hospital, Fudan University

IPD SHARING:
Plan to Share IPD: No